# **Protocol Clinical Trial (21/11/2018)**

#### Title of project

Blood eosinophil measurements in patients with Chronic Obstructive Pulmonary disease in stable state.

## **Objective**

To determine the within-day variation of blood eosinophils in patients with Chronic Obstructive Pulmonary disease in stable state.

To determine if there is a correlation between the blood eosinophils and certain clinical parameters.

# **Investigators**

I. Van Rossem, E. Vanderhelst, S. Hanon, S. Vincken, K. Jochmans, J. Vandevoorde

#### **Departments involved in the trial**

Department of Family Medicine and Chronic Care, Vrije Universiteit Brussel

Department of Internal Medicine, Division of Respiratory Disease, UZ Brussel

Department of Clinical Biology, UZ Brussel

# **Introduction**

Chronic Obstructive Pulmonary Disease (COPD) is a disease which leads to serious morbidity and mortality and it is currently the 4th leading cause of death in the world. (1) It is characterised by airflow limitation caused by a mixture of small airways disease and parenchymal destruction, the relative contributions of which vary from person to person. (2) It is a heterogeneous disease, resulting in different phenotypes with varying clinical and pathophysiological characteristics. One of these pathophysiological features is chronic airway inflammation and, although eosinophilic inflammation is thought to be a typical characteristic of asthma, there is mounting evidence that eosinophilic inflammation can also be present in COPD. (3)

Blood eosinophils are an accessible biomarker for the eosinophilic inflammation in COPD (3). Literature suggests a potential theragnostic role for this biomarker, seeing that COPD patients with higher levels of blood eosinophils could exhibit a greater responsiveness to corticosteroid treatments (4-7) and probably also to anti–IL-5 therapy. (8) Evidence also suggests that this biomarker could have a prognostic use for establishing the risk of exacerbations although conflicting results are found. (9)

But before being able to make decisions in the clinical management of patients based on blood eosinophils, more needs to be known about the different confounding factors and sources of within-subject variability of this biomarker. (10) As described by Brusselle et al. eosinophil counts can fluctuate due to their short half-life in blood and due to a diurnal rhythm. (11) There is evidence that this diurnal variation exists in healthy individuals (12) but, to the best of our knowledge, this has never been investigated in COPD patients before.

# Study design

Prospective interventional study

#### **Subjects**

Number and recruitment of subjects

50 COPD patients (GOLD A+B+C+D). All eligible COPD patients will be recruited at the respiratory unit of the UZ Brussel (included the patients admitted for nocturnal oximetry) or from family practices.

#### Inclusion criteria

Participant is willing and able to give informed consent for participation in the study. Patients are 18 years or older, with the diagnosis of COPD according to GOLD (post-bronchodilator Tiffeneau index <0.7), in stable state of the disease and with a smoking history of >10 pack-years.

#### Exclusion criteria

Clinical diagnosis of asthma

Use of systemic corticosteroids (oral, intravenous or infiltration up to six weeks before inclusion).

Pregnancy.

A recent exacerbation of COPD (<4 weeks ago).

#### Replacement of subjects

Inclusion of patients will continue until 50 patients have gone through the entire study protocol.

Restrictions and prohibitions for the subjects None.

#### **Procedures and collected variables**

Upon admission a questionnaire is filled in by the investigator or his representative: age, gender, smoking habits, weight, height, current medication, pulmonary function test with bronchodilation, mMRC (Modified Medical Research Council) Dyspnea Scale, exacerbation history in the previous year.

Fractional Exhaled Nictric Oxide (FENO) measurement and blood sampling at 08h00, 12h00, 16h00 (total red blood cell count, total white blood cell count with formula in absolute count and percentage of total white blood cells, and platelet count).

## **Randomisation/blinding**

Not applicable.

# **Prior and concomitant therapy**

Medication prohibited before and during the trial are systemic corticosteroids (oral, intravenous or infiltration, up to six weeks before inclusion). All other medication use is allowed.

## Study analysis

#### Sample size calculation

Due to the lack of previous research, a sample size calculation was impossible to perform and an arbitrary decision was made.

## Analysis of the samples

The analysis of the blood samples will be done at the Department of Clinical Biology, UZ Brussel. The pulmonary function test will be performed at the Department of Internal Medicine, Division of Respiratory Disease, UZ Brussel.

## Statistical analysis

Statistical analyses will be performed by the Department of Statistics and Data-analyses of the Vrije Universiteit Brussel.

#### **Quality control and quality assurance**

Quality control and quality assurance will be done according to guidelines of the Association for the Accreditation of Human Research Protection Programs.

#### **Data Protection**

## Responsible for processing of personal data

Department of Family Medicine and Chronic Care, Vrije Universiteit Brussel

Contact person: Inès Van Rossem, Vakgroep Huisartsgeneeskunde en Chronische Zorg, Vrije Universiteit Brussel, Laarbeeklaan 103, 1090 Jette, tel: +32 2 477 43 11

## Data Protection Officer (DPO)

Audrey van Scharen, DPO Vrije Universiteit Brussel (DPO@vub.be)

## Goal of the processing

The gathered data will be used for the academic scientific research purposes described in this protocol. It will be processed according to the principles imposed by the European General Data Protection Regulation (GDPR), which has been in force since 25 May 2018.

The legal basis for the processing is permission. There is an explicit permission from the data subject for the processing of personal data through informed consent. Permission can be withdrawn by the participant at any time, for any reason and without having to state a reason.

#### Recipients of data

The prime investigator and the study nurse will be the only individuals with access to personnel data. Study data will not be transferred to other countries.

## Storage

The study data will be stored in an excel file in a coded fashion with the encryption key held in a separate file. Both the data file and the encryption key will be password protected and saved in the one drive system of the Vrije Universiteit Brussel.

The gathered study data will be saved for a period of minimum 20 years. This in accordance with the Belgian law on experiments on the human person (7 May 2004).

## **Publication policy**

All authors will contribute to publication and hold all publication rights.

## **Funding**

A request for funding was submitted to the "Belgische Vereniging voor Pneumologie".

#### References

- 1. Lozano R, Naghavi M, Foreman K, et al. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet 2012; 380: 2095-2128.
- 2. Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2018. Available from: http://goldcopd.org.
- 3. Singh D, Kolsum U, Brightling CE et al. Eosinophilic inflammation in COPD: prevalence and clinical characteristics. Eur Respir J 2014; 44: 1697–1700.
- 4. Brightling CE, McKenna S, Hargadon B, et al. Sputum eosinophilia and the short term response to inhaled mometasone in chronic obstructive pulmonary disease. Thorax 2005; 60: 193–198.
- 5. Brightling CE, Monteiro W, Ward R, et al. Sputum eosinophilia and short-term response to prednisolone in chronic obstructive pulmonary disease: a randomised controlled trial. Lancet 2000; 356: 1480–1485.
- 6. Leigh R, Pizzichini MM, Morris MM, et al. Stable COPD: predicting benefit from high-dose inhaled corticosteroid treatment. Eur Respir J 2006; 27: 964–971.
- 7. Pizzichini E, Pizzichini MM, Gibson P, et al. Sputum eosinophilia predicts benefit from prednisone in smokers with chronic obstructive bronchitis. Am J Respir Crit Care Med 1998; 158: 1511–1517.
- 8. Pavord ID, Chanez P, Criner GJ, et al. Mepolizumab for eosinophilic chronic obstructive pulmonary disease. N Engl J Med 2017; 377: 1613–1629.
- 9. Vedel-Krogh S, Nielsen SF, Lange P, Vestbo J, Nordestgaard BG. Blood eosinophils and exacerbations in COPD: the Copenhagen General Populations Study. Am J Respir Crit Care Med 2016; 193: 965-974.
- 10. Gibson PG. Variability of blood eosinophils as a biomarker in asthma and COPD. Respirology 2018; 23: 12 –13.
- 11. Brusselle G, Pavord I, Landi S, et al. Blood eosinophil levels as a biomarker in COPD. Respir Med. 2018; 138: 21-31.
- 12. Winkel P, Statland BE, Saunders AM, Osborn H, Kupperman H. Within-day physiologic variation of leukocyte types in healthy subjects as assayed by two automated leukocyte differential analyzers. Am J Clin Pathol. 1981; 75: 693-700.

fautoseto

Dr. Inès Van Rossem